CLINICAL TRIAL: NCT01476956
Title: Prospective Validation of Soluble Biomarkers as Predictors of Structural Damage in Rheumatoid Arthritis
Brief Title: Assess Structural Damage in Rheumatoid Arthritis Using Biomarkers and Radiography
Status: Completed | Type: Observational
Sponsor: CARE ARTHRITIS LTD. (Industry)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: RA BIODAM
Record Dates: First submitted 2011-06-01; First posted 2011-11-22 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * whole blood/serum
  * urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — RA patients on standard DMARD therapy

SUMMARY:
Recruited patients will include those about to begin Disease-Modifying Antirheumatic Drug) DMARD therapy or about to change DMARD therapy.

Disease activity will be monitored systematically every 3 months by the Disease Activity Score.

Changes in standard DMARD and/or anti-Tumor Necrosis Factor α (anti-TNFα) therapy will be made according to specific recommendations for patients receiving these therapies.

Biomarker samples will be collected every 3 months and prior to change in DMARD and/or anti-TNF therapy as defined below. A blood sample (40 ml) for serum will be taken for biomarker studies and processed according to the international committee of Outcome Measures in Rheumatology (OMERACT) recommendations for the minimal handling of biomarker samples. A urine sample (20 ml) will also be taken and processed as for serum.

Radiography (X-rays) will be conducted every 6 months (baseline, 6, 12, 18, 24 months).

Patients will be followed for 2 years.

DETAILED DESCRIPTION:
Treatment is Disease Activity Score (DAS) driven. Changes in standard DMARD and/or anti-TNFα therapy will be implemented according to 2010 European League against Rheumatism (EULAR) recommendations which state a target of remission (DAS44 <1.6) for patients receiving standard DMARD therapy in the setting of early disease and a target of low disease activity state (LDAS) (DAS44 ≤2.4) for patients receiving anti-TNFα therapy in the setting of established disease.

ELIGIBILITY:
Inclusion Criteria (selected):

* 18 years of age or older
* RA according to the 2010 Rheumatoid Arthritis Classification Criteria
* Joint symptoms for ≥ 3 months prior to screening
* DAS44 > 2.4
* About to start DMARD therapy (methotrexate, salazopyrin, hydroxychloroquine, chloroquine, leflunomide) or

  * increased dose of methotrexate by ≥10 mg weekly to a maximum dose of 25mg weekly (if already receiving >15mg will require add-on DMARD/anti-TNF or switch to alternative DMARD),
  * add-on of alternative DMARD,
  * switch to alternative DMARD,
  * start of first anti-TNFα agent (adalimumab, etanercept, infliximab, certolizumab pegol, golimumab)
* If already on DMARD therapy this has been stable for the 3 months prior to the baseline visit
* If already on systemic steroid, dose must be stable (prednisone ≤ 7.5mg/day) for 1 month prior to the baseline visit
* Patient will be available for follow up for a minimum of 24 months from the baseline visit

Exclusion Criteria (selected):

* Intra-articular steroid injection within 4 weeks prior to the baseline visit
* Prior treatment with anti-TNFα or other biological agent (rituximab, abatacept, tocilizumab)
* Malignancy within past 5 years (other than basal cell carcinoma that has been adequately treated or excised, squamous cell cancer of the skin, and cervical carcinoma in situ)
* History of:

  * Serious infection (defined as requiring parenteral antibiotics or hospitalization) within 3 months prior to the baseline visit;
  * Active tuberculosis or history of tuberculosis without documented curative treatment and/or positive tuberculin reaction to PPD (Purified Protein Derivative)
* For patients starting anti-TNF therapy, a positive TB screening test and no record of effective prophylaxis according to local expert recommendations
* Known infection with Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patients from rheumatologists' clinics
Sampling Method: Non-Probability Sample
Enrollment: 571 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
To determine the independent predictive validity of several soluble biomarkers for predicting structural damage in Rheumatoid Arthritis (RA). | 24 Months

SECONDARY OUTCOMES:
To establish which modifiable clinical and laboratory predictors used in routine practice individually and in combination, have the strongest and the most consistent association with change in radiographic damage in patients on standard RA therapy. | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Walter P. Maksymowych, MD, Study Director — CaRE Arthritis
Locations (36):
- United States (5):
  - Johns Hopkins Arthritis Center, Johns Hopkins University, Baltimore, Maryland
  - Rheumatologist Hospital for Special Surgery, New York, New York
  - Division of Rheumatology, Columbia University, College of Physicians and Surgeons, New York, New York
  - Division of Allergy, Immunology and Rheumatology, University of Rochester, Rochester, New York
  - Seattle Rheumatology Associates, Seattle, Washington
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - Division of Rheumatology, University of Alberta Hospital, Edmonton, Alberta
  - Arthritis Center, University of Manitoba, Winnipeg, Manitoba
  - Memorial University, St. John's, Newfoundland and Labrador
  - The Arthritis Research Group, Newmarket, Ontario
  - University of Sherbrooke, Sherbrooke, Quebec
  - Saskatoon Osteoporosis Centre, Saskatoon, Saskatchewan
- Department of Rheumatology, Copenhagen University Hospital at Glostrup, Glostrup Municipality, Denmark
- France (6):
  - Service de Rheumatologie-CHU Bordeaux Pellegrin, Bordeaux
  - Le Roux Liana, Centre d'Investigation Clinique, Brest
  - Centre des Consultations et imagerie de l'appareil locomoteur service de rheumatologie, Lille
  - Departement de rheumatologie, Hopital Lapeyronie, Montpellier
  - Rheumatologie B, Hopital Cochin, Paris
  - Infirmiere de Recherche Clinique, CHU de Toulouse, Centre de Rheumatologie, Hopital Purpan, Toulouse
- Germany (4):
  - Kerckhoff-Klinik, Department of Rheumatology and Clinical Immunology, Bad Nauheim
  - Department of Rheumatology/Clinical Immunology, Medizinische Klinik-Rheumatologie und Klinische Immunologie, Berlin
  - Universitatsklinikum der Friedrich-Schiller-Universitat Jena, Klinik für Innere Medizin III/Rheumatologie/Osteologie, Jena
  - Dr Spieler, Zerbst
- Department of Rheumatology, St. Vincents University Hospital, Dublin, Ireland
- Tel Aviv Sourasky Medical Centre, Tel Aviv, Israel
- Italy (6):
  - University of Ferrara, Ferrara
  - University of Milan, Milan
  - Day Hospital Reumatologia, Milan
  - University of Padova, Padua
  - Catholic University of the Sacred Heart, Rome
  - Department of Rheumatology, University of Verona, Verona
- Netherlands (4):
  - Amsterdam VU University Medical Centre, Amsterdam
  - Academic Medical Centre/University of Amsterdam, Amsterdam
  - Academic Medical Centre/University of Amsterdam and Atrium Medical Centre Heerlen, Heerlen
  - Afdeling Reumatologie, Leids Universitair Medisch Centrum, Leiden
- Department of Rheumatology, Diakonhjemmet Hospital, Oslo, Norway

REFERENCES:
- [Derived] Sepriano A, Ramiro S, FitzGerald O, Ostergaard M, Homik J, van der Heijde D, Elkayam O, Thorne JC, Larche MJ, Ferraccioli G, Backhaus M, Burmester GR, Boire G, Combe B, Schaeverbeke T, Saraux A, Dougados M, Rossini M, Govoni M, Sinigaglia L, Cantagrel A, Barnabe C, Bingham CO 3rd, Tak PP, van Schaardenburg D, Hammer HB, Paschke J, Dadashova R, Hutchings E, Landewe R, Maksymowych WP. Adherence to Treat-to-target Management in Rheumatoid Arthritis and Associated Factors: Data from the International RA BIODAM Cohort. J Rheumatol. 2020 Jun 1;47(6):809-819. doi: 10.3899/jrheum.190303. Epub 2019 Sep 15. PMID 31523049
- [Derived] Maksymowych WP, FitzGerald O, Ostergaard M, Homik J, van der Heijde D, Lambert RG, Elkayam O, Ramiro S, Thorne JC, Larche MJ, Ferraccioli G, Backhaus M, Burmester GR, Boire G, Combe B, Schaeverbeke T, Saraux A, Dougados M, Rossini M, Govoni M, Sinigaglia L, Cantagrel A, Barnabe C, Bingham CO 3rd, Tak PP, van Schaardenburg D, Hammer HB, Paschke J, Dadashova R, Hutchings E, Sepriano A, Landewe R. Outcomes and Findings of the International Rheumatoid Arthritis (RA) BIODAM Cohort for Validation of Soluble Biomarkers in RA. J Rheumatol. 2020 Jun 1;47(6):796-808. doi: 10.3899/jrheum.190302. Epub 2019 Sep 1. PMID 31474600